CLINICAL TRIAL: NCT00110500
Title: A Phase I Dose-Escalation Clinical Trial of SB-509-0401 in Subjects With Diabetic Neuropathy
Brief Title: Clinical Trial of SB-509-0401 in Subjects With Diabetic Neuropathy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sangamo Therapeutics (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: SB-509-0401
Record Dates: First submitted 2005-05-09; First posted 2005-05-10 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-06

CONDITIONS: Diabetic Neuropathy
Keywords: Diabetes; Neuropathy
MeSH Terms: conditions — Diabetic Neuropathies; Diabetes Mellitus

INTERVENTIONS:
Genetic: hVEGF-A

SUMMARY:
The purpose of this study is to evaluate the clinical and laboratory safety of SB-509 when given as a single treatment by an intramuscular injection to subjects with diabetic neuropathy.

DETAILED DESCRIPTION:
Primary objective:

To evaluate the clinical and laboratory safety of SB-509 when given as a single treatment by an intramuscular injection. To determine the maximum tolerated dose (MTD) of a single treatment by intramuscular injection by SB-509.

Secondary objective:

To evaluate the lower extremity clinical effects of SB-509 treatment on lower limb diabetic neuropathy by symptoms, neurological examination, and lower extremity electrophysiological testing.

ELIGIBILITY:
Inclusion Criteria:

* Have a clinical diagnosis of Diabetes Mellitus Type I or II for at least 12 months prior to the study.
* Have received a diagnosis of mild to moderate sensori-motor diabetic neuropathy from a neurologist (a doctor who specializes in disorders of the nervous system) or endocrinologist (a doctor who specializes in diabetes). This type of neuropathy is a loss of sensation and muscle function that occurs in the legs and hands in a stocking and glove distribution. Subjects with diabetic neuropathy that results in loss of sensation or muscle function in only one nerve and results in loss of nerve function of the blood vessels and causes low blood pressure, will not be eligible.
* Be an adult male or female between the ages of 18 and 65.
* Be able and willing to read and sign a consent form.
* Be willing to participate in the study as an outpatient and make the required visits to the study center during the treatment and after the treatment periods
* Meet and follow the study requirements.
* Have abnormal signs of sensori-motor diabetic neuropathy based on a rating scale that is based on questions and a physical exam called the Neuropathy Impairment Score-Lower Limb (NIS-LL) clinical scoring system.
* Have abnormal results on specialized nerve testing in the legs. The study doctor or study staff will do this specialized nerve testing with a Nerve Conduction Test and Quantitative Sensory Testing, both of which you will read about below.
* Have measurable sural nerve responses in both legs
* Have an HgbA1C level that is 10% or lower, with stable blood sugar control for at least 3 months. The study doctor will check this.
* Have an eye exam by an eye doctor to rule out the presence of abnormal growth of blood vessels or proliferative diabetic retinopathy (eye complications of diabetes).
* Have a normal, complete blood count. The study doctor will check this.
* Have a normal urine test.
* If female, be: (a) postmenopausal or (b) surgically sterile or (c) use two forms of birth control and have a negative pregnancy test within 3 days of receiving the study drug.
* If male and able to make a female pregnant, use an accepted form of birth control.
* Have had up-to-date screening tests for cancer as recommended by the American Cancer Society. These tests include a PSA blood test for prostate cancer (for males over age 45), a pap smear for cervical cancer (for females), a mammogram (for females over age 40), and a flexible sigmoidoscopy for colon cancer (if over age 50). To be in this study, you must have written proof of normal test results within the last 12 months. If these screening tests show you have cancer, you will not be able to be in the study.
* Have a normal chest X-ray without evidence of heart enlargement or congestive heart failure.

Exclusion Criteria:

Subjects with the following are NOT eligible to participate in this study:

* Have moderate to severe ischemic heart disease, any history of congestive heart failure or have had a myocardial infarction (heart attack) within the previous 6 months.
* Have chronic foot or leg ulcers for >1 month, gangrene in the lower extremity, or any previous amputation of the lower extremity.
* Have symptoms of intermittent claudication (or leg pain during exercise associated with peripheral artery disease) and/or an ankle brachial index (or a calculation of the difference between arm and leg blood pressures) of less than < 0.75.
* Have a history of cancer within the past 10 years (except curable non-melanoma cancer of the skin, superficial bladder cancer in complete remission, or any other cancer that has been in complete remission for at least 5 years).
* Be pregnant, breastfeeding, or a man or woman of reproductive potential (able to make babies) not using an accepted form of birth control.
* Expect to require any surgery within 4 weeks of receiving the study drug.
* Have a condition that increases your risk of bleeding (for example, hemophilia or a similar disorder) or requires treatment with warfarin, clopidogrel, or aspirin (at least 325 mg each day) within 2 weeks before you receive the study drug and within 24 hours afterwards.
* Have had a stroke with bleeding in the brain within the last 12 months.
* Have had bleeding from the gastrointestinal tract (esophagus, stomach, duodenum, intestines, rectum) within the last 12 months. If you have ever had bleeding from the large intestine or rectum, you will need to have had a negative colonoscopy after that episode and within the last 3 years.
* Have any other condition that, in the opinion of the study doctor, might cause problems during the study (for example, affect your health or study test results).
* Be participating in another research study while you are in this study or within 30 days of receiving the study drug.
* Have colon polyps. If you have history of benign colonic polyps that have been removed, you must have evidence of a normal colonoscopy within the last 12 months.
* Have an inflammatory disorder of the blood vessels (inflammatory angiopathy, such as Buerger's disease).
* Have an active infection requiring antibiotics that you take by swallowing or is administered directly into a vein. If you had an infection in the past, you must not be receiving treatment for that infection within 2 weeks of receiving the study drug.
* Have abnormal kidney function.
* Require any drug that depresses your immune system (such as methotrexate, cyclophosphamide, or cyclosporine) when you receive the study drug and for 30 days afterwards.
* Have a known disorder that affects your immune system (such as HIV/AIDS, HBV, HCV, sarcoidosis, tuberculosis, rheumatoid arthritis, or autoimmune disorders).
* Be using oral, injectable, or intravenous (directly into the vein) corticosteroids (such as prednisone) within 30 days of starting the study.
* Have a history of drug addiction (not including smoking) within 12 months of the start of the study.
* Have any psychiatric (mental) or addictive disorders that would prevent the subject from being able to read and sign a consent form.
* Have neuropathy of the extremities that is caused by a condition other than diabetes (for example, alcohol abuse and liver or renal disease).
* Have received gene transfer agents within the last 6 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2005-04; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
To evaluate the clinical and laboratory safety of SB-509 when given as a single treatment by an intramuscular injection
To determine the maximum tolerated dose (MTD) of a single treatment by intramuscular injection by SB-509.

SECONDARY OUTCOMES:
To evaluate the lower extremity clinical effects of SB-509 treatment on lower limb diabetic neuropathy by symptoms, neurological examination, and lower extremity electrophysiological testing.

CONTACTS AND LOCATIONS:
Locations (1):
- San Antonio, Texas, United States

REFERENCES:
- See also: Sangamo Biosciences website — http://www.Sangamo.com